CLINICAL TRIAL: NCT04926792
Title: Taiwan Registry for Leadless Pacemaker
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taiwan Society of Cardiology (Unknown); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202103105RINB
Record Dates: First submitted 2021-06-09; First posted 2021-06-15 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Sick Sinus Syndrome; Atrioventricular Block
Keywords: Leadless Pacemaker; Taiwan
MeSH Terms: conditions — Sick Sinus Syndrome; Atrioventricular Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Leadless Pacemaker — Leadless pacemaker implantation

SUMMARY:
Taiwan Registry for Leadless Pacemaker is a nationwide registry for leadless pacemaker performance in Taiwan.

DETAILED DESCRIPTION:
The purpose of this registry is to investigate the safety and efficiency performance of the leadless pacemakers in Taiwan. The registry will collect all the information about the patient selection, implantation procedure, and follow up parameters of the leadless pacemakers to evaluate the real-world benefit specifically in Taiwan population.

ELIGIBILITY:
Inclusion Criteria:

1. The patients who had successfully received leadless pacemaker implantation
2. The patients who attempt to receive leadless pacemaker implantation

Exclusion Criteria:

N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: who attempt or had successfully received a leadless pacemaker implantation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute complication | On the 1 day of implant procedure
  Any acute complication during procedure
Subacute complication | within 3 month after implant procedure
  Any subacute complication, including pacemaker syndrome
Leadless Pacemaker performance | aroung 12 months after implant proceure
  The AV synchrony or pacemaker parameters

SECONDARY OUTCOMES:
Successful implant | 1 day
  The attempts of deployment in one procedure

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chieh Yu, MD.PhD, Principal Investigator — Taiwan Society of Cardiology
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No